CLINICAL TRIAL: NCT00800228
Title: Inhibited Breathing Pattern and Sodium Inhibitors in Sodium Sensitivity of Blood Pressure
Brief Title: Salt Study: Inhibited Breathing Pattern and Sodium Inhibitors in Sodium Sensitivity of Blood Pressure
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: David Anderson, Ph.D., National Institute on Aging, NIH
Other Study IDs: AG0110
Record Dates: First submitted 2008-11-30; First posted 2008-12-02 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-11

CONDITIONS: Hypertension
Keywords: salt; blood pressure; breathing
MeSH Terms: conditions — Hypertension; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Eight men and eight women to define the time course of changes in MBG \ and OLC accompanying sodium loading
- 2: 32 additional women to determine whether breathing pattern is predictive of sodium sensitivity in that gender. Women are being studied in the second experiment because they, but not men, have been shown to have an association of breathing pattern with high perceived stress11 and an association of high resting end tidal CO2 with high resting blood pressure.

SUMMARY:
The purpose of this study is to test the hypothesis that blood pressure sensitivity to high sodium intake in healthy humans is characterized by increased urinary excretion of two endogenous sodium pump inhibitors, marinobufagenin (MBG), and ouabain-like compound (OLC). The study also tests the hypothesis that women who breathe slowly and have high resting end tidal CO2 at rest are more likely to have low plasma renin activity and sodium sensitivity of blood pressure than those who breathe more rapidly and maintain lower end tidal CO2.

DETAILED DESCRIPTION:
The experiments will involve a common procedure of sodium restriction followed by sodium loading of normotensive (having normal blood pressure) humans. However, the first experiment will involve continuous urine collection throughout the experimental period in a smaller group of men and women, while the second experiment will involve urine collection only at the end of each diet period in a larger group of normotensive women. If, as expected, experiment one shows that sodium loading produces MBG increases that are sustained throughout the sodium loading period, then experiment two will also be able to address a third issue: that is whether MBG or OLC response to sodium loading is specific to breathing pattern or sodium sensitivity. It is hypothesized that women with inhibited breathing who are sodium sensitive will show higher levels of MBG, even before sodium loading, but also following sodium loading.

Each participant will be seen at the Clinical Research Unit for a screening visit and on days 6 and 12, and consume a low sodium diet for 6 days followed by a high sodium diet for 6 days. Research staff will meet with the participant at regular intervals for meal provision and transfer of 24-hr urine collections (if applicable). Respiration and blood pressure will be measured on the last day of each sodium diet.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70
* Caucasian
* Nonsmoking
* Free of respiratory, cardiac, liver and kidney disease, and diabetes
* Resting systolic blood pressure less than or equal to 139 mmHg AND resting diastolic blood pressure of less than or equal to 89 mmHg15
* BMI less than or equal to 30
* Negative pregnancy test for female participants whose last menstrual period was less than one year prior to study enrollment
* For Group 1, willing to provide 24-hr urine samples for 12 consecutive days
* For Group 2, women on combination oral contraceptives (those containing estrogen and progesterone) will be eligible for the study, with equal numbers in the "fast" and "slow" breathing groups
* For Group 2, in premenopausal women, regular menstrual cycles for at least 6 months prior to study entry

Exclusion Criteria:

* Presence of respiratory, cardiac, liver or kidney disease; diabetes, or hypertension
* Use of medications which can affect respiratory rate, such as major tranquilizers, narcotics, or benzodiazepines
* Diuretic or steroid use
* Cigarette smoking within the past 12 months
* BMI > 30 kg/m2
* Postmenopausal women on hormone replacement therapy
* Pregnancy or lactation in the last 12 months
* In premenopausal women, irregular menstrual cycles in the 6 months prior to study entry
* For Group 2, respiratory rate in the middle third of the distribution of breathing frequency in BLSA
* For Group 2, pre-menopausal women not taking oral contraceptives who are in the follicular phase of the menstrual cycle

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2003-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The sodium loading procedures will be identical in both experiments, except that 24-hr urine collection will be collected all 12 days in experiment one, but only on the last two days of each sodium diet in experiment two. | Group 1- daily; Group 2 - days 6 & 12

CONTACTS AND LOCATIONS:
Overall Officials: David Anderson, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- NIA Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Muntzel M, Drueke T. A comprehensive review of the salt and blood pressure relationship. Am J Hypertens. 1992 Apr;5(4 Pt 1):1S-42S. doi: 10.1093/ajh/5.4s.1s. PMID 1599633
- [Background] Haddy FJ. Digitalislike circulating factor in hypertension: potential messenger between salt balance and intracellular sodium. Cardiovasc Drugs Ther. 1990 Mar;4 Suppl 2:343-9. doi: 10.1007/BF02603174. PMID 2176807
- [Background] Doris PA, Bagrov AY. Endogenous sodium pump inhibitors and blood pressure regulation: an update on recent progress. Proc Soc Exp Biol Med. 1998 Jul;218(3):156-67. doi: 10.3181/00379727-218-44283. PMID 9648933
- [Background] Fedorova OV, Anderson DE, Lakatta EG, Bagrov AY. Interaction of NaCl and behavioral stress on endogenous sodium pump ligands in rats. Am J Physiol Regul Integr Comp Physiol. 2001 Jul;281(1):R352-8. doi: 10.1152/ajpregu.2001.281.1.R352. PMID 11404312